CLINICAL TRIAL: NCT03726541
Title: Hemodynamic Effects of Physiotherapy in the Early Postoperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Hemodynamics_ physiotherapy
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Physiotherapy; Postoperative; Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early physiotherapy group (Experimental): breathing exercise incentive spirometry training ambulation coughing
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — Physiotherapy program includes breathing exercises, incisive spirometer study, grade ambulation. Oxygen saturation, heart rate and blood pressure values will be recorded before and after the session. Changes in the follow-up parameters will be discussed.

SUMMARY:
Physiotherapy will be applied to the patients who undergo thoracotomy operation after 24 hours of intensive care stay. Physiotherapy program includes breathing exercises, incentive spirometer training, ambulation. Oxygen saturation, heart rate and blood pressure values will be recorded before and after the training session. Changes in the follow-up parameters will be discussed.

ELIGIBILITY:
Inclusion Criteria

* Between 18-75 age
* Hemodynamically stable
* Being conscious

Exclusion Criteria:

* Excessive pain
* Neurological complications
* Posttraumatic and musculoskeletal problems to prevent exercise
* Do not want to be included in the study
* Fever above 38 degrees

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline oxygen saturation | 30 minutes
  The hearth rate response will be measured before and after exercise training with pulse oximeter.
Change from baseline hearth rate response. | 30 minutes
  The hearth rate response will be measured before and after exercise training with intensive care ECG
Change from baseline systolic and diastolic blood pressure response. | 30 minutes
  Blood pressure will be measured before and after exercise training with monometer from the arm

CONTACTS AND LOCATIONS:
Overall Officials: Arif Balcı, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided